CLINICAL TRIAL: NCT03284229
Title: A Prospective, Open Label, Non-randomized, Single-Arm, Multicenter Study to Evaluate the Procedural Safety and Efficacy of ELCA® in Treatment of Patients With Single or Multivessel Coronary Artery Disease (CAD)
Brief Title: Multicenter Study to Evaluate the Procedural Safety and Efficacy of ELCA in CAD
Acronym: ELCA-CAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Spectranetics Corporation (Industry)
Collaborators: CBCC-VIBGYOR Research Pvt. Ltd. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ELCA-1016
Record Dates: First submitted 2017-09-08; First posted 2017-09-15 (Actual); Results first posted 2020-09-18 (Actual); Last update posted 2020-09-18 (Actual); Status verified 2020-07

CONDITIONS: Coronary Artery Disease
Keywords: ELCA; Coronary Artery Disease; India
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: As per the 25th SEC (Cardiovascular & Renal) meeting which deliberated the proposals on 30-10-2015 and recommended the firm (Spectranetics Corporation - Sponsor) shall conduct a Bridging study in Indian Population at least 25 patients with coronary artery disease. The directorate suggested that the sponsor submit a protocol for the study in India for clinical trial approval. Considering the 5 dropouts, Sponsor has set up this protocol to conduct the Excimer Laser Coronary Atherectomy (ELCA®) study in India on 30 eligible patients across 05 sites as a Stand-alone modality or in conjunction with Percutaneous Transluminal Coronary Balloon Angioplasty (PTCA) in single or multi-vessel coronary artery disease.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Excimer Laser Coronary Atherectomy (Experimental): ELCA® in patients with single or multivessel CAD either as a stand-alone modality or in conjunction with Percutaneous Transluminal Coronary Balloon Angioplasty (PTCA). The entire procedure will be carried out as per the site routine practice and the device will be used as per the 'Instruction for Use'. Treating physicians/study investigators will be trained by the study Sponsor on the study protocol and procedures prior to clinical investigation procedure. Subject preparation and percutaneous access should be performed according to the standard hospital practice. Both femoral and radial accesses are accepted.
  Interventions: Device: Excimer Laser Coronary Atherectomy

INTERVENTIONS:
Device: Excimer Laser Coronary Atherectomy — Excimer Laser Coronary Atherectomy (ELCA ®) uses the high energy, monochromatic light beam to alter or dissolve (vaporize) the plaque without damaging the surrounding tissue. Fiber-optic catheters are used to deliver this light beam. For endovascular applications, Xenon Chloride excimer laser is used and its fiber-optic catheter has multiple small fibers, rather than just a few large fibers, in order to be flexible enough to navigate in the arterial tree.
  Other Names: ELCA Coronary Laser Atherectomy Catheters (OTW and RX)

SUMMARY:
This is a Prospective, Open label, Non-randomized, Single-Arm, Multicenter Study to Evaluate the Procedural Safety and Efficacy of ELCA® in Treatment of Patients with Single or Multivessel Coronary Artery Disease (CAD). Up to 30 patients will be enrolled at up to 05 Indian study sites. Patients will be followed from enrollment through 30 days ± 7 days for the effectiveness and safety endpoints at the study centre.

DETAILED DESCRIPTION:
Each subject will be followed from enrollment through 30 days ± 7 days for the effectiveness and safety endpoints. Upon enrollment after obtaining a written informed consent, each patient will be assigned a unique identification number. Only patients eligible to undergo cardiac catheterizations as per routine practice will be considered for the study. Premedication of patients will be as per the investigator's routine practice. All patient data will be recorded on patient data forms.

Screening: This will be performed prior to the cardiac catheterization procedure. Only patients who have consented and fulfill the selection criteria will be enrolled. Additionally, ECG and Echocardiogram will be done using hospital equipment to ensure fulfillment of inclusion/exclusion criteria.

Procedure: The entire procedure will be carried out as per the site routine practice and the device will be used as per the IFU.

Clinic follow up visit (30 ± 7 days): The subject will return to the clinic at 1 month to evaluate angina status as per the CCS classification, AE assessments, concomitant medications and any coronary intervention that has occurred since the previous contact.

An electrocardiogram (ECG) will be repeated during the clinic visit.

ELIGIBILITY:
Inclusion Criteria:

* Have at least one severely stenotic lesion (greater than or equal to 80% diameter stenosis as assessed by visual estimation)
* Haemodynamically stable patients coming to the site for cardiac catheterization and angiography for various indications and who fulfill all the following criteria:
* Have no clinically significant cardiac arrhythmias, based on ECG results
* Have no evidence of valvular pathology, based on echocardiogram results
* Have ≥30% left ventricular ejection fraction (LVEF), based on echocardiogram results.
* Angiographic evidence of calcification or a chronic total occlusion
* Vessel reference diameter greater than or equal to 2.0 mm
* Patient is willing and able to comply with study requirements
* Women of child bearing potential, willing to use at least two methods of contraception

Exclusion Criteria:

* Evidence of acute coronary syndrome within 3 months prior to index procedure
* Evidence of acute ischemic events
* Cardiogenic and non-cardiogenic shock
* Active bleeding or coagulopathy
* Previous coronary angioplasty within 6 months of the index procedure
* Patients participating in trial for another investigational device/medicine within 1 month prior to enrolment in this study
* Acute or Chronic renal failure, Impaired renal function (serum creatinine > 2.5 mg/dl or 221 umol/l) determined within 72 hours prior to index procedure.
* Known allergies to the following: Aspirin, Clopidogrel or Ticlopidine, Heparin, Sirolimus or its derivatives, contrast agent (that cannot be adequately pre-medicated), or any metal
* Planned surgery within 6 months of enrollment in this study
* Life expectancy less than 6 months
* Patients known to be suffering from substance abuse (alcohol or drug)
* Patients with any other significant co-morbid illness which in the opinion of the investigator is not conducive of inclusion in the study.
* Known or suspected Pregnancy
* Patients not willing to provide written informed consent
* In the investigators opinion subjects will not be able to comply with the follow-up requirements.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2017-09-20 (Actual); Primary Completion 2018-05-21 (Actual); Study Completion 2018-05-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen Krygier, MBA, Study Director — Spectranetics Corporation
Locations (5):
- India (5):
  - Global Health Private Limited, Medanta - The Medicity, Gurgaon, Haryana
  - Sri Jayadeva Institute of Cardiovascular Sciences and Research, Bangalore, Karnataka
  - Lilavati Hospital and Research Centre, Bandra, Mumbai
  - Escorts Heart Institute & Research Centre Limited, New Delhi, National Capital Territory of Delhi
  - All Indian Institute of Medical Sciences (AIIMS), New Delhi, National Capital Territory of Delhi

REFERENCES:
- See also: ELCA laser system and catheter IFUs — http://www.spectranetics.com/resources/ifu-library/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 31 patients were screened. 3 patients were screen failure. 28 patients enrolled in the study.
Groups:
- Enrolled: Excimer Laser Coronary Atherectomy (ELCA) Enrolled Patients
Period: Overall Study
Arm/Group | Enrolled
Started | 28
Completed | 25
Not Completed | 3
Not completed — Lost to Follow-up | 3

BASELINE CHARACTERISTICS:
Groups:
- Enrolled: Enrolled Patients
Arm/Group | Enrolled
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.04 (8.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 19
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  India | 25
Height [Mean (Standard Deviation); unit: cms] — Height (cms)
  cms | 163.50 (8.68)
Weight [Mean (Standard Deviation); unit: kgs] — Weight (Kgs)
  kgs | 70.80 (11.37)
Angina Class [Count of Participants; unit: Participants] — Angina status or myocardial ischemia assessment as per the Canadian Cardiovascular Society (CCS) Classification.
  Grade I - ordinary physical activity does not cause angina. Angina with strenuous or rapid or prolonged exertion at work or recreation.
  Grade II - Slight limitation of ordinary activity. Grade III - Marked limitation of ordinary physical activity. Walking one or two blocks on the level and climbing one flight of stairs in normal conditions and at normal pace.
  Grade IV - Inability to carry on any physical activity without discomfort, anginal syndrome may be present at rest
  Participants
    Class 0/I | 3
    Class II | 17
    Class III | 4
    Class IV | 1

OUTCOME MEASURES:

1. Primary Outcome: Participants With Device Success During Procedure Defined as the Successful Crossing of the Laser Catheter Across the Entire Length of the Stenotic Lesion
Description: Successful crossing of the Laser Catheter across the entire length of the stenotic lesion
Time Frame: Procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Enrolled
Number analyzed (Participants) | 25
Participants
  Success | 25
  Failure | 0

2. Primary Outcome: Participants With Procedural Success Defined as Target Lesions With Less Than 50% Residual Stenosis After Laser and Adjunctive Therapy During Procedure
Description: Target lesions with less than 50% residual stenosis after laser and adjunctive therapy.
Time Frame: Procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Enrolled
Number analyzed (Participants) | 25
Participants
  < 50% | 25
  ≥ 50% | 0

3. Primary Outcome: Safety Success - Participants With Freedom From Major Adverse Cardiac Events (MACE) Defined as Death, Non-Q-wave and Q-wave Myocardial Infarction (MI), Target Lesion Revascularization, Cardiac Tamponade and Life Threatening Arrhythmias
Description: Freedom from Major Adverse Cardiac Events (MACE) defined as Death, Non-Q-wave and Q-wave myocardial infarction (MI), Target Lesion Revascularization, Cardiac tamponade and life threatening arrhythmias.
Time Frame: 30 days
Population: Safety success includes 25 subjects that completed follow up and 3 subjects that were Lost To Follow Up
Measure: Count of Participants; unit: Participants
Groups:
- Enrolled: Enrolled Patients, including Lost To Follow Up
Arm/Group | Enrolled
Number analyzed (Participants) | 28
Participants
  Death | 0
  Non-Q-wave | 0
  Q-wave myocardial infarction | 0
  Target Lesion Revascularization | 0
  Cardiac Tamponade | 0
  Life threatening arrhythmias | 0
  No Major Adverse Cardiac Events | 28

4. Secondary Outcome: TIMI Flow
Description: To determine post-procedural TIMI Flow grade. Changes of TIMI Grade flow after Index Procedure by measuring pre-procedure TIMI grade flow and post-procedure TIMI grade flow.
  TIMI flow is a scoring system from 0-3 referring to levels of coronary blood flow assessed during percutaneous coronary angioplasty. TIMI flow was assessed before and after the procedure. TIMI grade flow 0-3 are as described below.
  * TIMI 0 flow (no perfusion) refers to the absence of any antegrade flow beyond a coronary occlusion.
  * TIMI 1 flow (penetration without perfusion) is faint antegrade coronary flow beyond the occlusion, with incomplete filling of the distal coronary bed.
  * TIMI 2 flow (partial reperfusion) is delayed or sluggish antegrade flow with complete filling of the distal territory.
  * TIMI 3 is normal flow which fills the distal coronary bed completely.
Time Frame: pre-procedure and post-procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Enrolled
Number analyzed (Participants) | 25
Participants
  Pre-Procedure TIMI grade flow: TIMI grade flow 0 | 0
  Pre-Procedure TIMI grade flow: TIMI grade flow 1 | 12
  Pre-Procedure TIMI grade flow: TIMI grade flow 2 | 9
  Pre-Procedure TIMI grade flow: TIMI grade flow 3 | 4
  Post Procedure TIMI grade flow: TIMI grade flow 0 | 0
  Post Procedure TIMI grade flow: TIMI grade flow 1 | 0
  Post Procedure TIMI grade flow: TIMI grade flow 2 | 0
  Post Procedure TIMI grade flow: TIMI grade flow 3 | 25

5. Secondary Outcome: Lesion Morphology - Coronary Tortuosity Based on Degree of Tortuosity
Description: Tortuosity from coronary angiography
Time Frame: Procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Enrolled
Number analyzed (Participants) | 25
Participants
  < 45° | 14
  45° - 90° | 8
  > 90° | 3

6. Secondary Outcome: Lesion Morphology - Eccentricity of Coronary Lesion
Description: Eccentricity from coronary angiography as concentric (symmetric) or eccentric (asymmetric)
Time Frame: Procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Enrolled
Number analyzed (Participants) | 25
Participants
  Concentric lesions | 17
  Eccentric lesions | 8

7. Secondary Outcome: Lesion Morphology - Contour as a Lesion Characteristic
Description: Contour from coronary angiography
Time Frame: Procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Enrolled
Number analyzed (Participants) | 25
Participants
  Irregular Contour | 20
  Smooth Contour | 5

8. Secondary Outcome: Lesion Morphology - Bifurcation (Branch or Division of Artery)
Description: Bifurcation from coronary angiography
Time Frame: Procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Enrolled
Number analyzed (Participants) | 25
Participants
  Bifurcation | 0
  No Bifurcation | 25

9. Secondary Outcome: Participants With Device-related Complications During Procedure
Description: To determine device related complications
Time Frame: Procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Enrolled
Number analyzed (Participants) | 25
Participants
  Yes | 0
  No | 25

10. Secondary Outcome: Participants With Procedure-related Complications During Procedure
Description: To determine procedure related complications
Time Frame: Procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Enrolled
Number analyzed (Participants) | 25
Participants
  Yes | 0
  No | 25

ADVERSE EVENTS:
Time Frame: Adverse event data were collected throughout the clinical investigation in the case report form. Any adverse event will be followed until one month follow up visit.
Description: Adverse event definition and classification adapted from ISO 14155
Groups:
- Enrolled: Enrolled Patients, including LTFU
Arm/Group | Enrolled
All-Cause Mortality (participants affected / at risk) | 0/28
Serious Adverse Events (participants affected / at risk) | 0/28
Other Adverse Events (participants affected / at risk) | 3/28
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enrolled (N=28)
Cardiac troponin I increased (Investigations) | 1 (1)
Angina pectoris (Cardiac disorders) | 1 (1) — Stable angina pectoris
Dyspnoea exertional (Cardiac disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2016-10-12): https://cdn.clinicaltrials.gov/large-docs/29/NCT03284229/Prot_001.pdf